CLINICAL TRIAL: NCT07057206
Title: Simultaneous Engagement of Networks for Alleviating Pain (SENAP)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSU-2025-33913
Record Dates: First submitted 2025-06-13; First posted 2025-07-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neuropathic Pain; Postherpetic Neuralgia
Keywords: Neuropathic Pain; Post-Traumatic Pain; Post-Surgical Pain; Postherpetic Neuralgia; Central Pain Syndrome; Chronic Neuropathic Pain
MeSH Terms: conditions — Neuralgia; Neuralgia, Postherpetic; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PFM-guided cortical stimulation (Experimental): Abbott Eterna IPG and Lamitrode 44 paddles with accessory extensions and clinical programmers
  Interventions: Device: PFM-guided cortical stimulation

INTERVENTIONS:
Device: PFM-guided cortical stimulation — Abbott Eterna IPG and Lamitrode 44 paddles with accessory extensions and clinical programmers

SUMMARY:
This trial is investigating the acceptability and efficacy of PFM-guided cortical stimulation for the treatment of central neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years
* Clinical diagnosis of a refractory chronic neuropathic pain syndrome suggestive of deafferentation or central pain. Non-limiting examples of these syndromes are:
* post-traumatic pain syndromes (e.g. plexopathies, radiation-induced injury)
* postsurgical pain syndromes (e.g. phantom limb pain, anesthesia dolorosa)
* postherpetic neuralgia
* Central pain syndromes (e.g. post-stroke pain, multiple sclerosis pain, post-radiation pain)
* Greater than 6 months of chronic neuropathic pain
* Average pain intensity over the past 30 days reported as 6 or greater on a 0-10 numeric rating scale (NRS)
* Multidisciplinary pain consensus review that establishes
* Pain is refractory to medical management
* Pain that is refractory to or unlikely to be altered by less invasive treatment and
* Pain distribution either does not permit attempts at relief by a targeted nerve block (e.g., post-stroke pain) or such blocks have provided <25% relief.
* Medication doses currently stable (no active titration or drug trials in progress) in the 30 days prior to baseline (immediately pre-surgical) study visit
* Ability to speak / read English
* Capable of understanding and providing informed consent (verified if necessary by a standard tool such as the MacArthur Competency Assessment)
* Women of childbearing age must be on regular use of an accepted contraceptive method(s).

Exclusion Criteria:

* Pregnancy, breastfeeding, or unwilling to maintain regular use of contraceptives. Patients who become pregnant after enrollment may be excluded from the study if study procedures may cause risk to the fetus. Patients who become pregnant prior to the surgical implantation will be excluded from the study.
* Aphasia severe enough to limit the consent process or communication between the investigators and the patient. Patients with mild or recovering aphasia may be considered candidates at the discretion of the PI.
* Untreated or uncontrolled psychiatric illness (schizophrenia, bipolar disorder, obsessive-compulsive disorder), or personality disorders (e.g. borderline personality disorder) or other neuropsychiatric conditions that the evaluating clinician would recommend exclusion of the patient after neuropsychiatric evaluation.
* History of seizure disorder and seizure within the last year. Participants with a remote history of epilepsy will need documentation from their neurologist for eligibility.
* Suicide attempt within 12 months from baseline visit or imminent suicide risk in the judgment of study clinicians.
* Modified Scale for Suicidal Ideation Score of greater than or equal to 21
* History of diagnosed substance use disorder in the past 3 years. Benzodiazepines and/or opioids prescribed by a physician with use as directed do not count for this criterion. Cannabis/cannabinoid products will not be considered an exclusion if used under the auspices of a state-sponsored medical cannabis program.
* Major medical comorbidities increasing the risk of surgery including uncontrolled hypertension, severe diabetes, major organ system failure, need for chronic anticoagulation other than aspirin, active infection, immunocompromised state, or malignancy with < 5 years life expectancy.
* Inability to temporarily stop anticoagulation therapy (approximately 3 weeks total) for surgery and after surgery. Patients taking these medications will need to discuss the need/risk of continuing these medications with their physicians and the PI or study personnel may contact the treating physician(s) as well to discuss the risks of anticoagulation / antiaggregation therapy discontinuation.
* MRI (done within one year of the baseline period) with significant abnormalities other than those associated with the neurological disorder causing chronic pain.
* Implantable hardware not compatible with MRI or with the study or former metal worker that may pose risk from MRI.
* Previous ablative intracranial surgery for the management of a central pain syndrome.
* history of other neurosurgical procedures that may interfere with functioning of the device
* Active, pending, or planned litigation or workman's compensation claim related to the pain/injury. Current receipt of disability benefits, without a dispute or litigation, is not an exclusion.
* Requires ongoing or expected diathermy, electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) to treat a chronic condition
* Allergies or known hypersensitivity to materials in the implanted system (i.e. titanium, polyurethane, silicone, polyetherimide, stainless steel).
* Any other condition that, in the judgment of the PI or the Data Safety & Monitoring Board, significantly increases risk of receiving an implanted neurostimulator.
* Those who require ongoing monitoring of a disease state by MRI.
* Inability to target the somatocognitive action network or cingulate opercular network on fMRI

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 12 months
  Percentage of participants enrolled in the study who then undergo surgery and undergo externalized stimulation testing followed by implantation of the implantable pulse generator (IPG)

SECONDARY OUTCOMES:
NRS Pain Scale | 12 months
  Difference in numerical pain rating scale (NRS) between the best stimulation (sample of 5) and sham stimulation (sample of 5). Min-Max values: (0-10) where lower scores indicate a better outcome (more pain reduction)

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, Principal Investigator — University of Minnesota; Alexander Herman, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No